CLINICAL TRIAL: NCT02870413
Title: The Acceptability, Feasibility, and Impact of Telelactation Among Rural Mothers
Brief Title: Expanding Rural Access to Breastfeeding Support Via Telehealth: The Tele-MILC Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Lori Uscher-Pines, Policy Researcher, RAND
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2016-0194-AM03
Record Dates: First submitted 2016-08-10; First posted 2016-08-17 (Estimated); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Breastfeeding
Keywords: telehealth
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telelactation support (Experimental): Participants in the experimental group will receive unlimited, free telelactation visits with lactation consultants (IBCLCs) as demanded up to 12 weeks post-partum. Services will be available through mobile phone app.
  Interventions: Behavioral: Telelactation services
- Usual care (No Intervention): Participants in the control arm will receive care as usual.

INTERVENTIONS:
Behavioral: Telelactation services — Mothers will get unlimited access (for a three month period) to video calls with lactation consultants who are available 24/7. Mothers can use the service as demanded.
  Other Names: Virtual/remote breastfeeding support
  Arms: Telelactation support

SUMMARY:
The investigators will conduct a randomized controlled trial (RCT) to generate data on the impact of direct-to-consumer "telelactation" (virtual breastfeeding support) services. We will explore the feasibility, acceptability, and impact of these services. Postpartum mothers age 18 and older who have initiated breastfeeding will be recruited at a critical access hospital without access to IBCLCs in rural Pennsylvania and randomized into two study arms: 1) outpatient telelactation services via video calls on personal devices or 2) usual care. Data on breastfeeding duration and exclusivity, as well as perceptions and satisfaction with breastfeeding, will be captured via surveys and in-depth interviews and compared across groups.

DETAILED DESCRIPTION:
Increasing breastfeeding rates is an ongoing public health priority because of the health and economic benefits for infants, mothers, and communities. Professional lactation support, specifically by International Board Certified Lactation Consultants (IBCLCs), increases breastfeeding duration and exclusivity. Rural and underserved mothers have lower breastfeeding rates, and limited access to professional lactation support may contribute to this disparity. As such, the Surgeon General identifies increasing access to IBCLCs as a policy priority. Virtual "telelactation" consults that use two-way video have the potential to increase access to IBCLC services in rural settings that lack them. Several companies have begun to offer telelactation through a direct-to-consumer (DTC) model, where patients initiate video calls with providers using their personal devices including mobile phones, tablets, and laptops. While four studies with small samples explored the use of antiquated videoconferencing technology (i.e., that required dedicated equipment) for lactation support, no research has studied DTC telelactation or linked telelactation with breastfeeding outcomes. To address this evidence gap, the investigators will conduct a randomized controlled trial (RCT) to generate data on the feasibility, acceptability, and impact of DTC telelactation services. Postpartum mothers age 18 and older who have initiated breastfeeding will be recruited at a critical access hospital without access to IBCLCs in rural Pennsylvania and randomized into two study arms: 1) outpatient telelactation services via video calls on personal devices or 2) usual care. Data on breastfeeding duration and exclusivity, as well as perceptions and satisfaction with breastfeeding and with telelactation services, will be captured via surveys and in-depth interviews and compared across groups. This study will be the first experimental evaluation of telelactation and the first ever evaluation of DTC telelactation services. The results will inform policy debates about reimbursement and regulation of DTC telehealth services and the strengths and limitations of this model of healthcare delivery as applied to breastfeeding. It also has the potential to promote breastfeeding, one of the most widely recommended health behaviors among underserved families, and improve children's health in rural settings.

ELIGIBILITY:
Inclusion Criteria for mothers:

1. ≥ 18 years;
2. Initiated breastfeeding while in the hospital and intend to breastfeed post-discharge
3. Fluent in English

Inclusion criteria for infants:

1. Infants must be term or near term (>35 weeks gestational age)
2. Not require a stay in the neonatal intensive care unit

Exclusion Criteria:

1. Prisoners, incarcerated individuals, detainees, parolees, probationers will be excluded because there may external circumstances outside of their control that may prevent continuous breastfeeding.
2. Mothers and infants will be excluded if they have maternal, fetal, or neonatal conditions or complications with the potential to physiologically compromise breastfeeding or milk supply (e.g., infant cardiac defects, post-partum infant ventilator dependence), and or contraindications to breastfeeding as specified by the American Academy of Pediatrics (e.g., HIV+ status).

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 203 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Any breastfeeding (yes/no) at 3 months | Three months
Exclusive breastfeeding (yes/no) at 3 months | Three months

SECONDARY OUTCOMES:
Breastfeeding satisfaction (self-reported via questionnaire at 3 months postpartum) | Three months
  Survey question which captures extent of satisfaction with the experience of breastfeeding. Question reads: How satisfied do you feel about the experience of breastfeeding your baby over the past three months? (Very unsatisfied, somewhat unsatisfied, neither unsatisfied nor satisfied, somewhat satisfied, very satisfied). We will create a binary variable (satisfied vs. unsatisfied) based on this response, with those reporting "somewhat satisfied" or "very satisfied" defined as "satisfied."

CONTACTS AND LOCATIONS:
Locations (1):
- RAND Corporation, Arlington, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Uscher-Pines L, Ghosh-Dastidar B, Bogen DL, Ray KN, Demirci JR, Mehrotra A, Kapinos KA. Feasibility and Effectiveness of Telelactation Among Rural Breastfeeding Women. Acad Pediatr. 2020 Jul;20(5):652-659. doi: 10.1016/j.acap.2019.10.008. Epub 2019 Oct 16. PMID 31629118
- [Derived] Kapinos K, Kotzias V, Bogen D, Ray K, Demirci J, Rigas MA, Uscher-Pines L. The Use of and Experiences With Telelactation Among Rural Breastfeeding Mothers: Secondary Analysis of a Randomized Controlled Trial. J Med Internet Res. 2019 Sep 3;21(9):e13967. doi: 10.2196/13967. PMID 31482848